CLINICAL TRIAL: NCT04351438
Title: Prismaflex Therapeutic Plasma Exchange: Evaluation of Complication Rates Using Filter vs. Centrifuge and Heparin vs. Citrate Anticoagulation
Brief Title: Evaluation of Complication Rates Using Filter vs. Centrifuge and Heparin vs. Citrate Anticoagulation
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, David Askenazi, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: 300003769
Record Dates: First submitted 2020-04-10; First posted 2020-04-17 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Therapeutic Plasma Exchange; Anticoagulant Therapy
Keywords: complications; heparin; citrate; membrane; filter
MeSH Terms: interventions — Citric Acid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- Centrifuge TPE with citrate: These participants were undergoing centrifuge TPE using citrate anticoagulant
  Interventions: Device: Active Comparator: centrifuge TPE with citrate
- Filter TPE with heparin: These participants were undergoing filter TPE using filter-based heparin anticoagulant
  Interventions: Device: Active Comparator: Filter TPE with heparin
- Filter TPE with citrate: These participants were undergoing filter TPE using filter-based citrate anticoagulant
  Interventions: Drug: Active comparator: Filter TPE with citrate

INTERVENTIONS:
Device: Active Comparator: centrifuge TPE with citrate — Patients who received citrate-based anticoagulation with centrifuge TPE
  Groups: Centrifuge TPE with citrate
Device: Active Comparator: Filter TPE with heparin — Patients who received heparin-based anticoagulation with filter TPE
  Groups: Filter TPE with heparin
Drug: Active comparator: Filter TPE with citrate — Patients who received citrate-based anticoagulation with filter TPE
  Groups: Filter TPE with citrate

SUMMARY:
Despite its growing use across the world, and similar efficacy, filter-based therapeutic plasma exchange (TPE) continues to be used less often that centrifuge-based TPE. One of the reasons is that the patient and circuit complications of centrifuge-based TPE are familiar to the clinical team. There is little data on the patient and circuit complications of filter-based TPE (using the Prismaflex). Furthermore, there is a reluctance to use filter-based TPE because historically, most TPE programs have used citrate-regional anticoagulation, and there is a large gap in knowledge in the use of citrate regional anti-coagulation when using filter-based TPE.

DETAILED DESCRIPTION:
Studies that evaluate differences between filter-based vs. centrifuge based TPE are lacking. Heparin-based TPE is the most commonly used method of anti-coagulation when performing filter-based TPE. Citrate anticoagulation is FDA approved for use during TPE and its use is the gold-standard anti-coagulant method for TPE. However, citrate has not been studied rigorously in patients who are on filtration-based TPE on Prismaflex.

Providing citrate-based anticoagulation during TPE is challenging for several reasons. First, because calcium will bind to albumin, one must provide additional albumin in some way to prevent hypocalcemia. Second, when the replacement fluid is fresh frozen plasma (FFP), the clinician must account for a very large dose of citrate (which can be 3 times higher than the dose used to anti-coagulate whole blood) that is present in the FFP. Based on these principles, with clinical observations and experience using citrate-based continuous renal replacement therapy, this hospital developed a clinical protocol for use during filter-based TPE. This protocol has been in use since 2012 in the Renal Care Center at the Children's of Alabama.

As the use of filter-based TPE continue to rise, clinicians need evidence-based data to help them care for their patients. Although there are a few reports on the complication rates during centrifuge TPE, known, there are no published reports on the complication rate during filter-based TPE. A comparison of the complications rate between filter-based TPE and centrifuge TPE will help providers recognize the safety of filter-based TPE. There are no known regional citrate anticoagulation protocols for patients receiving filter-based TPE using Prismaflex. As the use of filter-based TPE continues to rise, there is a great need to fill this important knowledge gap. As more patients are cared in critical care arena, more clinicians will need evidence-based protocols for regional citrate anti-coagulation. This study will fill important gaps in knowledge that will improve the ability of clinical teams to provide filter-based TPE using Prismaflex.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received therapeutic plasma exchange at Children's of Alabama between 2012 and 2019

Exclusion Criteria:

* Patients that received TPE with concomitant extra-corporeal membrane oxygenation

Ages: 0 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: retrospective database used to analyze subjects
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2024-02-04 (Actual)

PRIMARY OUTCOMES:
Percentage of patient complications during TPE | complications during any TPE procedure (3 hours to 400 days)
  patient-related complications during procedure

SECONDARY OUTCOMES:
Percentage of circuit-related complications during TPE | 4 hours
  circuit-related complications during procedure

CONTACTS AND LOCATIONS:
Overall Officials: David Askenazi, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kellum JA, Lameire N; KDIGO AKI Guideline Work Group. Diagnosis, evaluation, and management of acute kidney injury: a KDIGO summary (Part 1). Crit Care. 2013 Feb 4;17(1):204. doi: 10.1186/cc11454. PMID 23394211
- [Result] Zhang W, Bai M, Yu Y, Li L, Zhao L, Sun S, Chen X. Safety and efficacy of regional citrate anticoagulation for continuous renal replacement therapy in liver failure patients: a systematic review and meta-analysis. Crit Care. 2019 Jan 24;23(1):22. doi: 10.1186/s13054-019-2317-9. PMID 30678706
- [Result] Meersch M, Kullmar M, Wempe C, Kindgen-Milles D, Kluge S, Slowinski T, Marx G, Gerss J, Zarbock A; SepNet Critical Care Trials Group. Regional citrate versus systemic heparin anticoagulation for continuous renal replacement therapy in critically ill patients with acute kidney injury (RICH) trial: study protocol for a multicentre, randomised controlled trial. BMJ Open. 2019 Jan 21;9(1):e024411. doi: 10.1136/bmjopen-2018-024411. PMID 30670518
- [Result] Zhang C, Lin T, Zhang J, Liang H, Di Y, Li N, Gao J, Wang W, Liu S, Wang Z, Jiang H, Liu C. [Safety and efficacy of regional citrate anticoagulation in continuous renal replacement therapy in the presence of acute kidney injury after hepatectomy]. Zhonghua Wei Zhong Bing Ji Jiu Yi Xue. 2018 Aug;30(8):777-782. doi: 10.3760/cma.j.issn.2095-4352.2018.08.013. Chinese. PMID 30220281
- [Result] Rico MP, Fernandez Sarmiento J, Rojas Velasquez AM, Gonzalez Chaparro LS, Gastelbondo Amaya R, Mulett Hoyos H, Tibaduiza D, Quintero Gomez AM. Regional citrate anticoagulation for continuous renal replacement therapy in children. Pediatr Nephrol. 2017 Apr;32(4):703-711. doi: 10.1007/s00467-016-3544-9. Epub 2016 Nov 28. PMID 27896442
- [Result] Lee G, Arepally GM. Anticoagulation techniques in apheresis: from heparin to citrate and beyond. J Clin Apher. 2012;27(3):117-25. doi: 10.1002/jca.21222. Epub 2012 Apr 24. PMID 22532037
- [Result] Kankirawatana S, Huang ST, Marques MB. Continuous infusion of calcium gluconate in 5% albumin is safe and prevents most hypocalcemic reactions during therapeutic plasma exchange. J Clin Apher. 2007;22(5):265-9. doi: 10.1002/jca.20142. PMID 17722047
- [Result] Lemaire A, Parquet N, Galicier L, Boutboul D, Bertinchamp R, Malphettes M, Dumas G, Mariotte E, Peraldi MN, Souppart V, Schlemmer B, Azoulay E, Canet E. Plasma exchange in the intensive care unit: Technical aspects and complications. J Clin Apher. 2017 Dec;32(6):405-412. doi: 10.1002/jca.21529. Epub 2017 Feb 1. PMID 28146331